CLINICAL TRIAL: NCT02547038
Title: Comparing the Efficacy and Impact on Gastrointestinal Microbiome of Reverse Hybrid Therapy and Bismuth Quadruple Therapy in Helicobacter Pylori Eradication
Brief Title: Comparing the Efficacy of Reverse Hybrid Therapy and Bismuth Quadruple Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Ping-I (William) Hsu, M.D., Professor, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: VGHKS15-CT2-10
Record Dates: First submitted 2015-09-06; First posted 2015-09-11 (Estimated); Results first posted 2019-06-10 (Actual); Last update posted 2019-06-10 (Actual); Status verified 2019-03

CONDITIONS: Helicobacter Pylori Infection
Keywords: Helicobacter pylori; Eradication rate
MeSH Terms: interventions — Pantoprazole; bismuth tripotassium dicitrate; Tetracycline; Metronidazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- pantoprazole+bismuth+tetra+metro (Experimental): pantoprazole 40 mg twice daily, bismuth subcitrate 120 mg four times daily, and tetracycline 500 mg four times daily, and metronidazole 250 mg four times daily for 14 days
  Interventions: Drug: pantoprazole+bismuth+tetra+metro
- (panto+amox+clar+metr)+(panto+amox) (Active Comparator): a 7-day quadruple regimen with pantoprazole 40 mg twice daily, amoxicillin 1 g twice daily, clarithromycin 500 mg twice daily, and metronidazole 500 mg twice daily, followed by a 7-day dual regimen with pantoprazole 40 mg twice daily and amoxicillin 1 g twice daily
  Interventions: Drug: (panto+amox+clar+metr)+(panto+amox)

INTERVENTIONS:
Drug: pantoprazole+bismuth+tetra+metro — pantoprazole 40 mg twice daily, bismuth subcitrate 120 mg four times daily, and tetracycline 500 mg four times daily, and metronidazole 250 mg four times daily for 14 days
  Other Names: pantoprazole 40 mg; bismuth subcitrate 120 mg; tetracycline 500 mg; metronidazole 250 mg
  Arms: pantoprazole+bismuth+tetra+metro
Drug: (panto+amox+clar+metr)+(panto+amox) — a 7-day quadruple regimen with pantoprazole 40 mg twice daily, amoxicillin 1 g twice daily, clarithromycin 500 mg twice daily, and metronidazole 500 mg twice daily, followed by a 7-day dual regimen with pantoprazole 40 mg twice daily and amoxicillin 1 g twice daily
  Other Names: pantoprazole 40 mg; amoxicillin 1 g; clarithromycin 500 mg; metronidazole 500 mg
  Arms: (panto+amox+clar+metr)+(panto+amox)

SUMMARY:
Reverse hybrid therapy achieves a higher eradication rate than bismuth quadruple therapy remained unanswered.

DETAILED DESCRIPTION:
A 14-day hybrid therapy invented by our study group appears very promising in H. pylori eradication, achieving excellent eradication rates of 99% and 97% according to per-protocol and intention-to-treat analyses, respectively. Recently, the investigators demonstrated that the eradication rate of reverse hybrid therapy was higher than that of standard triple therapy. However, whether reverse hybrid therapy achieves a higher eradication rate than bismuth quadruple therapy remained unanswered.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive H pylori-infected outpatients, at least 20 years of age, with endoscopically proven peptic ulcer diseases or gastritis

Exclusion Criteria:

* previous H pylori-eradication therapy
* ingestion of antibiotics or bismuth within the prior 4 weeks
* patients with allergic history to the medications used
* patients with previous gastric surgery
* the coexistence of serious concomitant illness (for example, decompensated liver cirrhosis, uremia)
* pregnant women

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2015-02; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ping-I Hsu, Bachelor, Study Chair — Kaohsiung Veterans General Hospital.
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

REFERENCES:
- [Background] Vakil N, Megraud F. Eradication therapy for Helicobacter pylori. Gastroenterology. 2007 Sep;133(3):985-1001. doi: 10.1053/j.gastro.2007.07.008. PMID 17854602
- [Background] Hunt RH, Lam SK. Helicobacter pylori: from art to a science. J Gastroenterol Hepatol. 1998 Jan;13(1):21-8. doi: 10.1111/j.1440-1746.1998.tb00540.x. PMID 9737567
- [Background] Fock KM, Katelaris P, Sugano K, Ang TL, Hunt R, Talley NJ, Lam SK, Xiao SD, Tan HJ, Wu CY, Jung HC, Hoang BH, Kachintorn U, Goh KL, Chiba T, Rani AA; Second Asia-Pacific Conference. Second Asia-Pacific Consensus Guidelines for Helicobacter pylori infection. J Gastroenterol Hepatol. 2009 Oct;24(10):1587-600. doi: 10.1111/j.1440-1746.2009.05982.x. PMID 19788600
- [Background] Asaka M, Kato M, Takahashi S, Fukuda Y, Sugiyama T, Ota H, Uemura N, Murakami K, Satoh K, Sugano K; Japanese Society for Helicobacter Research. Guidelines for the management of Helicobacter pylori infection in Japan: 2009 revised edition. Helicobacter. 2010 Feb;15(1):1-20. doi: 10.1111/j.1523-5378.2009.00738.x. PMID 20302585
- [Background] Malfertheiner P, Megraud F, O'Morain CA, Atherton J, Axon AT, Bazzoli F, Gensini GF, Gisbert JP, Graham DY, Rokkas T, El-Omar EM, Kuipers EJ; European Helicobacter Study Group. Management of Helicobacter pylori infection--the Maastricht IV/ Florence Consensus Report. Gut. 2012 May;61(5):646-64. doi: 10.1136/gutjnl-2012-302084. PMID 22491499
- [Background] Chey WD, Wong BC; Practice Parameters Committee of the American College of Gastroenterology. American College of Gastroenterology guideline on the management of Helicobacter pylori infection. Am J Gastroenterol. 2007 Aug;102(8):1808-25. doi: 10.1111/j.1572-0241.2007.01393.x. Epub 2007 Jun 29. PMID 17608775
- [Background] Graham DY, Shiotani A. New concepts of resistance in the treatment of Helicobacter pylori infections. Nat Clin Pract Gastroenterol Hepatol. 2008 Jun;5(6):321-31. doi: 10.1038/ncpgasthep1138. Epub 2008 Apr 29. PMID 18446147
- [Background] Megraud F. H pylori antibiotic resistance: prevalence, importance, and advances in testing. Gut. 2004 Sep;53(9):1374-84. doi: 10.1136/gut.2003.022111. No abstract available. PMID 15306603
- [Background] Luther J, Higgins PD, Schoenfeld PS, Moayyedi P, Vakil N, Chey WD. Empiric quadruple vs. triple therapy for primary treatment of Helicobacter pylori infection: Systematic review and meta-analysis of efficacy and tolerability. Am J Gastroenterol. 2010 Jan;105(1):65-73. doi: 10.1038/ajg.2009.508. Epub 2009 Sep 15. PMID 19755966
- [Background] De Francesco V, Margiotta M, Zullo A, Hassan C, Troiani L, Burattini O, Stella F, Di Leo A, Russo F, Marangi S, Monno R, Stoppino V, Morini S, Panella C, Ierardi E. Clarithromycin-resistant genotypes and eradication of Helicobacter pylori. Ann Intern Med. 2006 Jan 17;144(2):94-100. doi: 10.7326/0003-4819-144-2-200601170-00006. PMID 16418408
- [Background] Gumurdulu Y, Serin E, Ozer B, Kayaselcuk F, Ozsahin K, Cosar AM, Gursoy M, Gur G, Yilmaz U, Boyacioglu S. Low eradication rate of Helicobacter pylori with triple 7-14 days and quadriple therapy in Turkey. World J Gastroenterol. 2004 Mar 1;10(5):668-71. doi: 10.3748/wjg.v10.i5.668. PMID 14991935
- [Background] Bigard MA, Delchier JC, Riachi G, Thibault P, Barthelemy P. One-week triple therapy using omeprazole, amoxycillin and clarithromycin for the eradication of Helicobacter pylori in patients with non-ulcer dyspepsia: influence of dosage of omeprazole and clarithromycin. Aliment Pharmacol Ther. 1998 Apr;12(4):383-8. doi: 10.1046/j.1365-2036.1998.00315.x. PMID 9690730
- [Background] De Francesco V, Margiotta M, Zullo A, Hassan C, Giorgio F, Burattini O, Stoppino G, Cea U, Pace A, Zotti M, Morini S, Panella C, Ierardi E. Prevalence of primary clarithromycin resistance in Helicobacter pylori strains over a 15 year period in Italy. J Antimicrob Chemother. 2007 Apr;59(4):783-5. doi: 10.1093/jac/dkm005. Epub 2007 Feb 28. PMID 17329269
- [Background] Zullo A, De Francesco V, Hassan C, Morini S, Vaira D. The sequential therapy regimen for Helicobacter pylori eradication: a pooled-data analysis. Gut. 2007 Oct;56(10):1353-7. doi: 10.1136/gut.2007.125658. Epub 2007 Jun 12. PMID 17566020
- [Background] Essa AS, Kramer JR, Graham DY, Treiber G. Meta-analysis: four-drug, three-antibiotic, non-bismuth-containing "concomitant therapy" versus triple therapy for Helicobacter pylori eradication. Helicobacter. 2009 Apr;14(2):109-18. doi: 10.1111/j.1523-5378.2009.00671.x. PMID 19298338
- [Background] Hsu PI, Wu DC, Wu JY, Graham DY. Modified sequential Helicobacter pylori therapy: proton pump inhibitor and amoxicillin for 14 days with clarithromycin and metronidazole added as a quadruple (hybrid) therapy for the final 7 days. Helicobacter. 2011 Apr;16(2):139-45. doi: 10.1111/j.1523-5378.2011.00828.x. PMID 21435092
- [Background] Malfertheiner P, Bazzoli F, Delchier JC, Celinski K, Giguere M, Riviere M, Megraud F; Pylera Study Group. Helicobacter pylori eradication with a capsule containing bismuth subcitrate potassium, metronidazole, and tetracycline given with omeprazole versus clarithromycin-based triple therapy: a randomised, open-label, non-inferiority, phase 3 trial. Lancet. 2011 Mar 12;377(9769):905-13. doi: 10.1016/S0140-6736(11)60020-2. Epub 2011 Feb 21. PMID 21345487
- [Background] Sardarian H, Fakheri H, Hosseini V, Taghvaei T, Maleki I, Mokhtare M. Comparison of hybrid and sequential therapies for Helicobacter pylori eradication in Iran: a prospective randomized trial. Helicobacter. 2013 Apr;18(2):129-34. doi: 10.1111/hel.12017. Epub 2012 Nov 4. PMID 23121338
- [Background] Zullo A, Scaccianoce G, De Francesco V, Ruggiero V, D'Ambrosio P, Castorani L, Bonfrate L, Vannella L, Hassan C, Portincasa P. Concomitant, sequential, and hybrid therapy for H. pylori eradication: a pilot study. Clin Res Hepatol Gastroenterol. 2013 Dec;37(6):647-50. doi: 10.1016/j.clinre.2013.04.003. Epub 2013 Jun 6. PMID 23747131
- [Background] De Francesco V, Hassan C, Ridola L, Giorgio F, Ierardi E, Zullo A. Sequential, concomitant and hybrid first-line therapies for Helicobacter pylori eradication: a prospective randomized study. J Med Microbiol. 2014 May;63(Pt 5):748-752. doi: 10.1099/jmm.0.072322-0. Epub 2014 Feb 28. PMID 24586031
- [Background] Oh DH, Lee DH, Kang KK, Park YS, Shin CM, Kim N, Yoon H, Hwang JH, Jeoung SH, Kim JW, Jang ES, Jung HC. Efficacy of hybrid therapy as first-line regimen for Helicobacter pylori infection compared with sequential therapy. J Gastroenterol Hepatol. 2014 Jun;29(6):1171-6. doi: 10.1111/jgh.12518. PMID 24955448
- [Background] Wang B, Wang YH, Lv ZF, Xiong HF, Wang H, Yang Y, Xie Y. Review: efficacy and safety of hybrid therapy for Helicobacter pylori infection: a systematic review and meta-analysis. Helicobacter. 2015 Apr;20(2):79-88. doi: 10.1111/hel.12180. Epub 2014 Nov 8. PMID 25381839
- [Background] Molina-Infante J, Romano M, Fernandez-Bermejo M, Federico A, Gravina AG, Pozzati L, Garcia-Abadia E, Vinagre-Rodriguez G, Martinez-Alcala C, Hernandez-Alonso M, Miranda A, Iovene MR, Pazos-Pacheco C, Gisbert JP. Optimized nonbismuth quadruple therapies cure most patients with Helicobacter pylori infection in populations with high rates of antibiotic resistance. Gastroenterology. 2013 Jul;145(1):121-128.e1. doi: 10.1053/j.gastro.2013.03.050. Epub 2013 Apr 3. PMID 23562754
- [Background] Chuah SK, Tsay FW, Hsu PI, Wu DC. A new look at anti-Helicobacter pylori therapy. World J Gastroenterol. 2011 Sep 21;17(35):3971-5. doi: 10.3748/wjg.v17.i35.3971. PMID 22046084
- [Background] Georgopoulos SD, Papastergiou V, Karatapanis S. Helicobacter pylori Eradication Therapies in the Era of Increasing Antibiotic Resistance: A Paradigm Shift to Improved Efficacy. Gastroenterol Res Pract. 2012;2012:757926. doi: 10.1155/2012/757926. Epub 2012 Jun 19. PMID 22778723
- [Background] Rimbara E, Fischbach LA, Graham DY. Optimal therapy for Helicobacter pylori infections. Nat Rev Gastroenterol Hepatol. 2011 Feb;8(2):79-88. doi: 10.1038/nrgastro.2010.210. PMID 21293508
- [Background] Wu DC, Hsu PI, Wu JY, Opekun AR, Kuo CH, Wu IC, Wang SS, Chen A, Hung WC, Graham DY. Sequential and concomitant therapy with four drugs is equally effective for eradication of H pylori infection. Clin Gastroenterol Hepatol. 2010 Jan;8(1):36-41.e1. doi: 10.1016/j.cgh.2009.09.030. Epub 2009 Oct 3. PMID 19804842
- [Background] Hsu PI, Lai KH, Tseng HH, Liu YC, Yen MY, Lin CK, Lo GH, Huang RL, Huang JS, Cheng JS, Huang WK, Ger LP, Chen W, Hsu PN. Correlation of serum immunoglobulin G Helicobacter pylori antibody titers with histologic and endoscopic findings in patients with dyspepsia. J Clin Gastroenterol. 1997 Dec;25(4):587-91. doi: 10.1097/00004836-199712000-00007. PMID 9451668
- [Background] Hsu PI, Wu DC, Chen A, Peng NJ, Tseng HH, Tsay FW, Lo GH, Lu CY, Yu FJ, Lai KH. Quadruple rescue therapy for Helicobacter pylori infection after two treatment failures. Eur J Clin Invest. 2008 Jun;38(6):404-9. doi: 10.1111/j.1365-2362.2008.01951.x. Epub 2008 Apr 22. PMID 18435764
- [Background] Hsu PI, Wu DC, Chen WC, Tseng HH, Yu HC, Wang HM, Kao SS, Lai KH, Chen A, Tsay FW. Randomized controlled trial comparing 7-day triple, 10-day sequential, and 7-day concomitant therapies for Helicobacter pylori infection. Antimicrob Agents Chemother. 2014 Oct;58(10):5936-42. doi: 10.1128/AAC.02922-14. Epub 2014 Jul 28. PMID 25070099
- [Background] Peng NJ, Lai KH, Liu RS, Lee SC, Tsay DG, Lo CC, Tseng HH, Huang WK, Lo GH, Hsu PI. Clinical significance of oral urease in diagnosis of Helicobacter pylori infection by [13C]urea breath test. Dig Dis Sci. 2001 Aug;46(8):1772-8. doi: 10.1023/a:1010626225949. PMID 11508681
- [Derived] Hsu PI, Tsay FW, Graham DY, Tsai TJ, Tsai KW, Kao JY, Peng NJ, Kuo CH, Kao SS, Wang HM, Lin TF, Wu DC; Taiwan Acid-related Disease (TARD) Study Group. Equivalent Efficacies of Reverse Hybrid and Bismuth Quadruple Therapies in Eradication of Helicobacter pylori Infection in a Randomized Controlled Trial. Clin Gastroenterol Hepatol. 2018 Sep;16(9):1427-1433. doi: 10.1016/j.cgh.2018.03.031. Epub 2018 Mar 31. PMID 29609070

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruitment period: August 2015 through February 2017. Type of location: Kaohsiung Veterans General Hospital and Kaohsiung Medical University Chung-Ho Memorial Hospital
Pre-assignment Details: None were excluded following participant enrollment.
Period: Overall Study
Arm/Group | Pantoprazole+Bismuth+Tetra+Metro | (Panto+Amox+Clar+Metr)+(Panto+Amox)
Started | 176 | 176
Completed | 173 | 174
Not Completed | 3 | 2
Not completed — Lost to Follow-up | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pantoprazole+Bismuth+Tetra+Metro | (Panto+Amox+Clar+Metr)+(Panto+Amox) | Total
Number analyzed (Participants) | 176 | 176 | 352
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 145 | 137 | 282
  >=65 years | 31 | 39 | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.8 (12.1) | 54.5 (12.9) | 54.2 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 97 | 87 | 184
  Male | 79 | 89 | 168
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 176 | 176 | 352
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 176 | 176 | 352
History of smoking [Number; unit: participants] | 24 | 35 | 59

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Which H. Pylori Was Eradicated
Description: Evaluate eradication outcome by endoscopy urease test and histology or urea breath test (Number of Participants With Complete Eradication of Helicobacter Pylori)
Time Frame: sixth week after the end of anti- H. pylori therapy
Population: Intention to treat
Measure: Number; unit: participants
Arm/Group | Pantoprazole+Bismuth+Tetra+Metro | (Panto+Amox+Clar+Metr)+(Panto+Amox)
Number analyzed (Participants) | 176 | 176
participants | 169 | 170

ADVERSE EVENTS:
Time Frame: 2 months
Arm/Group | Pantoprazole+Bismuth+Tetra+Metro | (Panto+Amox+Clar+Metr)+(Panto+Amox)
All-Cause Mortality (participants affected / at risk) | 0/176 | 0/176
Serious Adverse Events (participants affected / at risk) | 0/176 | 0/176
Other Adverse Events (participants affected / at risk) | 86/176 | 33/176
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pantoprazole+Bismuth+Tetra+Metro (N=176) | (Panto+Amox+Clar+Metr)+(Panto+Amox) (N=176)
Nausea (General disorders) | 67 (67) | 15 (15) — Patients had Nausea discomforts.
Dizziness (General disorders) | 13 (13) | 4 (4) — Patients had dizziness discomforts.
Abdominal pain (Gastrointestinal disorders) | 5 (5) | 7 (7) — Patients had dizziness discomforts.
Diarrhea (Gastrointestinal disorders) | 1 (1) | 7 (7) — Patients had dizziness discomforts.

LIMITATIONS AND CAVEATS:
The trial was performed in a single country

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/38/NCT02547038/Prot_SAP_000.pdf